CLINICAL TRIAL: NCT06444464
Title: The BEE-Power Study (Boosting Exercise for Excellent Pediatric Blood Pressure)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 276902; P20GM109096 (NIH)
Record Dates: First submitted 2024-05-23; First posted 2024-06-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Overweight and Obesity; Adolescent Obesity; Exercise
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Active Comparator): After baseline 24-hour blood pressure measurements are taken at visit 2, participants will attend a final study visit where they will engage in a single session of aerobic exercise. The exercise routines will include 5 to 10-minute warm-up and cool-down periods, along with a 30-minute workout. Twenty-four hour blood pressure measurements will be taken after the exercise bout.
  Interventions: Other: Aerobic exercise
- Isometric Exercise (Experimental): After baseline 24-hour blood pressure measurements are taken at visit 2, participants will attend a final study visit where they will engage in a single session of isometric exercise. The exercise routines will include 5 to 10-minute warm-up and cool-down periods, along with a 30-minute workout. Twenty-four hour blood pressure measurements will be taken after the exercise bout.
  Interventions: Other: Isometric exercise

INTERVENTIONS:
Other: Aerobic exercise — After baseline 24-hour blood pressure measurements are taken at visit 2, participants will attend a final study visit where they will engage in a single session of aerobic exercise. The exercise routines will include 5 to 10-minute warm-up and cool-down periods, along with a 30-minute workout. Twenty-four hour blood pressure measurements will be taken after the exercise bout.
  Arms: Aerobic Exercise
Other: Isometric exercise — After baseline 24-hour blood pressure measurements are taken at visit 2, participants will attend a final study visit where they will engage in a single session of isometric exercise. The exercise routines will include 5 to 10-minute warm-up and cool-down periods, along with a 30-minute workout. Twenty-four hour blood pressure measurements will be taken after the exercise bout.
  Arms: Isometric Exercise

SUMMARY:
The goal of this study is to compare two types of exercises, isometric exercise (like squats and planks) and aerobic exercise (such as running), to see which one is more effective at improving blood pressure in teenagers aged 13 to 17.5 years.

The main question the study aims to answer is:

- Do the effects of one session of isometric exercise on the blood pressure of adolescents compare to the effects of one session of aerobic exercise?

Adolescents with overweight or obesity may qualify for this study. Participants will be randomly assigned to either a single session of isometric exercise or a single session of aerobic exercise.

* Participants will attend 3 study visits in total.
* Study visits should be completed within 4 weeks of enrollment.
* At the initial visit, samples (example: blood) will be collected and body measurements will be taken.
* Participants will be asked to answer questionnaires (diet, growth, and others)
* At visit 2, participants will have their blood pressure measured using a 24 hour blood pressure monitor.
* At visit 3, participants will participate in a single session of either aerobic or isometric exercise. They will wear a 24-hour blood pressure monitor immediately after the exercise session.

DETAILED DESCRIPTION:
Our approach to testing our working hypotheses will be to enroll children ages 13 to <18 years of age. Children will be divided equally into two groups (aerobic exercise and isometric exercise groups), with 18 children in each group. Children who meet inclusion criteria will be asked to attend three study visits at the Arkansas Children's Nutrition Center (ACNC). Resting and 24-hour ambulatory blood pressure measurements will be conducted twice during the study: baseline measurement at visit 2 and after a single session of exercise at visit 3. To accommodate for any potential dropouts post-assignment and to maintain an even distribution of participants between groups (n =18 each), the study will enroll up to n = 45 children (Refer to the Data Analysis and Randomization section for more details).

The study will follow a randomized parallel group design and will be conducted by the Physical Activity Core - Arkansas Children's Nutrition Center (ACNC) / Arkansas Children's Research Institute in collaboration with the Hypertension Clinic - Nephrology Division at the Arkansas Children Hospital (ACH). Measurements will be completed within four weeks of enrollment. Research staff involved in study procedures are or will be properly trained. All assessments may be repeated if/when needed, and if the participant is willing. Study visits may last up to 3 hours.

Baseline characteristics such as socioeconomic status, pubertal stage, dietary quality, physical fitness (aerobic capacity, body composition) and metabolic phenotyping (glucose, insulin, lipids, etc.) will be used to control for baseline covariates as described in the Data analysis Section.

ELIGIBILITY:
Inclusion Criteria

* Age 13 to less than 18 years old.
* Excessive weight: BMI percentile ≥ 85th percentile.

Exclusion Criteria

* Asthma that requires daily use of inhalers to keep symptoms under control
* Asthma that requires use of rescue inhalers (e.g., albuterol) >2 days per week
* Exercise induced asthma
* Autism spectrum disorder (e.g., Autistic disorder, Rett disorder, Asperger disorder, childhood disintegrative disorder, pervasive developmental disorder not otherwise specified (PDD-NOS)
* Attention deficit hyperactivity disorder (ADHD) treated with medication or unwillingness to discontinue medication 1 day prior to the study visit and during ambulatory blood pressure monitoring.
* Oppositional defiant disorder (ODD)
* Epilepsy
* Cancer
* Chronic kidney disease
* Autoimmune diseases (e.g., lupus, thyroiditis, juvenile idiopathic arthritis)
* Bleeding disorders (e.g., hemophilia)
* Chronic infections (e.g., HIV, hepatitis B, hepatitis C)
* Type 2 and type 1 diabetes mellitus.
* Other pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest.
* Parent/participant refusal to have blood drawn
* Unwillingness to wear a 24-hour ambulatory blood pressure monitor.
* Hypertension managed with medication
* Allergy to latex

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Mean (24-hour) systolic and diastolic blood pressure | Within 4 weeks after enrollment: at visits 2 and 3
  The 24-hour average of systolic and diastolic blood pressure will be calculated from data collected using ambulatory blood pressure monitoring.
Mean systolic and diastolic blood pressure during sleep | Within 4 weeks after enrollment: at visits 2 and 3
  The mean systolic and diastolic blood pressure during sleep will be calculated from data collected using ambulatory blood pressure monitoring.
Mean systolic and diastolic blood pressure during the awake period | Within 4 weeks after enrollment: at visits 2 and 3
  The mean systolic and diastolic blood pressure during the awake period will be calculated from data collected using ambulatory blood pressure monitoring.
Nocturnal dipping pattern | Within 4 weeks after enrollment: at visits 2 and 3
  Nocturnal dipping pattern will be calculated as follows: Percent day- night BP difference

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Diaz, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No